CLINICAL TRIAL: NCT03413709
Title: New Pathways to Responsible Fatherhood Family Formation Program
Brief Title: Fathers' Support Center New Pathways to Responsible Fatherhood Family Formation Program (NPFF) Impact Evaluation Plan
Acronym: NPFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fathers' Support Center, St. Louis (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Cheri Tillis, Project Director, Fathers' Support Center, St. Louis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201605068
Record Dates: First submitted 2016-09-28; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Parenting
Keywords: Parenting Time, Father Involvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (n=350) (Active Comparator): The sample for the treatment group for the impact evaluation will only include fathers who are receiving the full 240 hour Family Formation Program (and not the abbreviated 80 hour program). The treatment group will receive FSC's Family Formation Program, which is a six week, 240 hour program implementing a set of curricula focusing on responsible parenting, healthy relationships,and economic stability and mobility. In addition, participants will receive case management and a variety of employment, legal and support services for up to one year following the completion of the curriculum.
  Interventions: Other: Family Formation Program
- Comparison Group (n=350) (No Intervention): The sample comparison group will receive only the abbreviated 80 hour program. Which consist of economic stability and mobility only. These participants will receive employment case management and legal services for up to one year following the completion of the curriculum.

INTERVENTIONS:
Other: Family Formation Program — The sample for the treatment group for the impact evaluation will only include fathers who are receiving the full 240 hour FFP program (and not the abbreviated 80 hour program). The treatment group will receive FSC's Family Formation Program, which is a six week, 240 hour program implementing a set of curricula focusing on responsible parenting, healthy relationships, and economic stability and mobility.
  Other Names: Economic Stability; Health Relationships; Responsible Parenting
  Arms: Treatment Group (n=350)

SUMMARY:
The Fathers' Support Center, in partnership with the Brown School Evaluation Center at Washington University in St. Louis, seeks to evaluate the impact of their New Pathways to Responsible Fatherhood Family Formation Program (NPFF). The investigators are most interested in quantifying the added benefit of parenting, father-child engagement, and father well-being curriculum compared to course content containing 80 hour economic stability material only. The impact evaluation will answer four key outcome and implementation specific questions using a mixed methods approach. Participants will be randomly assigned to one of two groups (full program or 80 hour economic stability curriculum only) and tracked for the duration of the program. The impact evaluation tools include a set of validated instruments and will be administered to participants at baseline and again at three and twelve months after completion of the program. Performance measurement data will also be included in our analysis. Investigators hypothesize that participation in the full program will have a greater effect on key outcomes than the economic stability curriculum, a similar number of families will be reached by each condition, and that there will be minimal variability in retention rates across groups.

DETAILED DESCRIPTION:
Research Questions

The Brown School Evaluation Center at Washington University in St. Louis will conduct the local impact evaluation. The local evaluation seeks to answer four primary questions pertaining to the implementation and outcomes of the Family Formation Program (FFP) (an integrated approach of responsible parenting, economic stability and mobility, and healthy relationships):

Outcome Q1: Does the participation of fathers in the comprehensive Family Formation Program have greater effect on family functioning, father and child outcomes, and father economic stability and mobility compared to fathers receiving the 80 hour economic stability services only (i.e., job readiness and employment skills)?

Implementation Q2: How many families were reached by each of the conditions and was there variability in retention rates of fathers across conditions?

Implementation Q3: Did fathers in the treatment and comparison conditions find the intervention to be acceptable and appropriate?

Implementation Q4: What barriers and benefits exist to successful implementation of father focused family support programs?

Background Fatherhood programs originally had a narrow focus on financial stability and support, but have recently evolved to also emphasize healthy relationships, parenting skills, and father involvement. Despite significant state and federal funding for fatherhood programs, few have undergone rigorous evaluation to examine their effectiveness. This evaluation will determine the added benefit of content on parenting, father-child engagement, and father well-being over and above content on economic stability and mobility, in relation to family functioning, child well-being, and economic stability. This will also further build the evidence supporting one particular comprehensive intervention, FFP, as a means to improve outcomes for children and families through intervening with fathers.

Relation to program logic model The primary research question of this impact evaluation will examine the effect of the FFP on short- and long-term outcomes as described in the FFP logic model

Short-term outcomes assessed by the impact evaluation will include:

1. improved parenting and co-parenting skills;
2. increased father-child engagement;
3. increased financial responsibility of fathers; and
4. progress towards greater economic stability.

The impact evaluation will also examine the FFP long-term outcomes of improved family functioning (through changes in father and child well-being; co-parenting relationship quality, and the father-child relationship) and increased economic stability and mobility.

Hypothesis:

Investigators believe that the FFP will have a greater effect on family functioning, father and child outcomes, and father economic stability compared to fathers in the comparison group because members of the treatment group will be receiving a more comprehensive range of services. Investigators anticipate that fathers will equally participate in both programs because both will provide meaningful information and opportunities to build their skill sets.

ELIGIBILITY:
Inclusion Criteria:

* being a father (biological or step) with at least one child 16 years old or younger

Exclusion Criteria:

* no presence of a restraining order from mother or child
* is not currently incarcerated
* is not homeless

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Father Engagement-Father Research & Practice Network (FRPN) Father Engagement Scale | 1 year from program completion
  Brief instrument designed to assess fathers' engagement with children at different ages. Separate scales for fathers of children ages 0-1 years, 1-5 years, 6-12 years, and adolescents. Scales found to have good reliability and validity
Father Child Contact-nForm Survey | 1 year from program completion
  Pre- and post-program nForm survey items related to father-child contact will be used to evaluate this construct.
Child Behavior and Emotion-Child Behavior Checklist (CBCL) | 1 year from program completion
  Standardized instrument based on national norms that assesses child behavioral and emotional problems. Study will use anxious/depressed and aggressive behavior sub-scales.
Parental Health-SF12v2 Health Survey | 1 year from program completion
  12-item nationally-normed health survey that measures functional health and well-being from the patient's point of view.
Parental Substance Abuse-Alcohol Use Disorder Identification Test (AUDIT) | 1 year from program completion
  10-item screening tool developed by World Health Organization to assess alcohol use, alcohol dependence, and alcohol-related problems. Its reliability and validity have been established in research conducted in a variety of settings
Parental Consequences related to Drug Abuse-Drug Abuse Screening Test 10 (DAST-10) | 1 year from program completion
  Brief instrument that yields a quantitative index of the degree of consequences related to drug abuse. Literature has shown moderate to high reliability and validity
Parental Discipline Strategies/Behavior-Conflict Tactics Scale-Parent Child (CTSPC) | 1 year from program completion
  Well-established instrument used to assess physical and psychological maltreatment. Study will use minor assault and non-violent discipline sub-scale items only
Co-parenting Relationships-FRPN: Coparenting Relationship Scale | 1 year after completion
  11-item measure designed to assess fathers' coparenting relationships with the mother of their children. The measure was validated with a sample of fathers very similar to those served in U.S. responsible fatherhood programs
Child/Financial Support Behavior-FSC Intake Survey | 1 year after program completion
  Items from FSC intake survey related to child and financial support will be used to assess this construct.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Green, Study Chair — Washington University, Human Research Protection Office
Locations (1):
- Fathers Support Center, St. Louis INC., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kohl PL, Krauss MJ, King C, Cheng SY, Fowler P, Goodwin DN, Tillis CD, Sullivan H, Sorg A, Mueller NB. The impact of responsible fatherhood programs on parenting, psychological well-being, and financial outcomes: A randomized controlled trial. Fam Process. 2022 Sep;61(3):1097-1115. doi: 10.1111/famp.12752. Epub 2022 Jan 5. PMID 34988991